CLINICAL TRIAL: NCT01097083
Title: A Randomized Phase II Trial of Coriolus Versicolor as Palliative Therapy Compared to Placebo in Patients With Child-Pugh C Unresectable Hepatocellular Carcinoma or Who Are Unfit for Standard Therapy
Brief Title: Coriolus Versicolor as Palliative Therapy Compared to Placebo in Patients With Child-Pugh C Unresectable Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2010-03-30; First posted 2010-04-01 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Carcinoma; Therapy
Keywords: Patients With Child-Pugh C Unresectable Hepatocellular Carcinoma; Patients who are unfit for standard therapy
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Coriolus Versicolor

SUMMARY:
The hypothesis of this study is that the median time to progression in the experimental arm is 2 months as compared to the placebo arm of 1.4 months

ELIGIBILITY:
Inclusion Criteria:

The diagnosis of HCC is made either by histological examination of tumor tissue or imaging evidence of a typical space-occupying lesion in the liver together with a serum AFP concentration of above 500 ng/ml (normal value, 10 ng/ml) in a known carrier of hepatitis B or C, or AFP above 400 ng/ml in non Hepatitis B or C carrier.

* Patients with unresectable HCC that is not amenable to liver transplantation nor local ablative technique and who are not suitable for any conventional systemic therapy (including sorafenib and chemotherapy).
* Patients with Child-Pugh Class C liver cirrhosis (Child-Pugh Scores of 10-15 points). Patients with Child-Pugh Class A or B liver cirrhosis who are not eligible for conventional therapy or other clinical trials or who refuse conventional therapy are included
* Life Expectancy of at least 12 weeks
* All patients should have anti-HBc antibodies tested if HBs Ag is negative. If anti-HBc is positive, HBV DNA detection should be performed to determine viral load. An undetectable Hep B DNA level (DNA levels < 12 IU/ml) in the presence of a positive Hep B core total antibody would indicate no active hepatitis infection and the subject would still be eligible for this trial.
* Age >21 years.
* Performance status ECOG 0 - 2
* Patients must have normal organ and marrow function as defined below:

Absolute neutrophil count > 1.5 x 109/L Platelets > 50 x 109/L Haemoglobin > 9.0g/dl Total bilirubin < 51umol/L (3 mg /dL) AST (SGOT)/ALT (SGPT) < 5 X institutional ULN Creatinine < 1.5 ULN INR <1.7 or prothrombin time (PT) <4 seconds above ULN

* Patients who have not received any local or systemic treatment in the last 4 weeks.
* Measurable disease according to RECIST
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow oral medication
* The effects of C versicolor on the developing human fetus are unknown. For this reason, woman of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Patients with a history of prior malignancy that is distinct in site and histology from HCC except non-melanoma skin cancer. Any cancer curatively treated more than 3 years prior to entry is permitted.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, intractable ascites that could not be controlled by medical therapy
* Prior use of C versicolor or Yunzhi for HCC
* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who are using other chinese herbal therapies concurrently or on any other investigation agents for treatment of their cancer
* Known of history of allergic reactions attributed to compounds of similar chemical or biologic composition used in the study.
* Presence of active hepatitis B/C flare.
* Known history of Human Immunodeficiency Virus (HIV) Infection
* Gastrointestinal disease which could affect the absorption or pharmacokinetics of the study drug as determined by investigator
* Psychiatric illness/social situations that would limit compliance with study requirements. Patients with severe depression or psychiatric disorders will be excluded.
* Known alcohol and/or substance abuser that may interfere with the subject's participation in the study or evaluation of study results.
* Pregnancy or breast-feeding subjects. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) within the 14 days prior to study enrollment and must be willing to use adequate contraception
* Patients suffering from autoimmune disease, patients on concomitant long-term immunosuppressant therapy and those scheduled to receive bone marrow transplants

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2010-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Peng Yong, MRCP, MB ChB', Principal Investigator — National University Hospital, Singapore; Choo Su Pin, BMBS, MRCP, M Med, Principal Investigator — National Cancer Centre; Tan Chee Kiat, MBBS, FRCP, FAMS, Principal Investigator — Singapore General Hospital
Locations (3):
- Singapore (3):
  - National University Hospital, Singapore, Singapore
  - Singapore General Hospital, Singapore
  - National Cancer Centre, Singapore

REFERENCES:
- [Background] Okuda K, Ohtsuki T, Obata H, Tomimatsu M, Okazaki N, Hasegawa H, Nakajima Y, Ohnishi K. Natural history of hepatocellular carcinoma and prognosis in relation to treatment. Study of 850 patients. Cancer. 1985 Aug 15;56(4):918-28. doi: 10.1002/1097-0142(19850815)56:43.0.co;2-e. PMID 2990661
- [Background] Falkson G, Ryan LM, Johnson LA, Simson IW, Coetzer BJ, Carbone PP, Creech RH, Schutt AJ. A random phase II study of mitoxantrone and cisplatin in patients with hepatocellular carcinoma. An ECOG study. Cancer. 1987 Nov 1;60(9):2141-5. doi: 10.1002/1097-0142(19871101)60:93.0.co;2-4. PMID 2830952